CLINICAL TRIAL: NCT00737867
Title: Vinorelbine Plus Gemcitabine (VG) Versus Vinorelbine Plus Carboplatin (VC) in Advanced Non-small Cell Lung Cancer. An Open Randomized Multicenter Phase III Trial From Norwegian Lung Cancer Study Group (NLCG)
Brief Title: Vinorelbine/Gemcitabine Versus Vinorelbine/Carboplatin in Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Norwegian Lung Cancer Study Group (Network)
Responsible Party: Øystein Fløtten, Haukeland University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11066741577; Eudra-CT-nr 2006-002927-18
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-04

CONDITIONS: Advanced Non-Small Cell Lung Cancer
Keywords: lung cancer; chemotherapy; vinorelbine; gemcitabine; carboplatin; advanced lung cancer; non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Vinorelbine; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Day 1: Vinorelbine (Navelbine® Oral) capsules 60 mg/m2 + Gemcitabine infusion 1000 mg/m2 Day 8: Vinorelbine (Navelbine® Oral) capsules 60 mg/m2 + Gemcitabine infusion 1000 mg/m2
  All patients will receive a maximum of 3 courses with an interval of 3 weeks
  Interventions: Drug: Vinorelbine; Drug: Gemcitabine
- B (Active Comparator): Day 1: Vinorelbine (Navelbine® Oral) capsules 60 mg/m2 + Carboplatin infusion AUC = 5 (Calvert's formula) Day 8: Vinorelbine (Navelbine® Oral) capsules 60 mg/m2
  All patients will receive a maximum of 3 courses with an interval of 3 weeks
  Interventions: Drug: Vinorelbine; Drug: Carboplatin

INTERVENTIONS:
Drug: Vinorelbine — Day 1: Vinorelbine capsules 60 mg/m2 Day 8: Vinorelbine capsules 60 mg/m2
  Other Names: Navelbine® Oral
  Arms: A
Drug: Gemcitabine — Day 1: Gemcitabine infusion 1000 mg/m2 Day 8: Gemcitabine infusion 1000 mg/m2
  Other Names: Gemzar; Gemcitabin
  Arms: A
Drug: Vinorelbine — Day 1: Vinorelbine capsules 60 mg/m2 Day 8: Vinorelbine capsules 60 mg/m2
  Other Names: Navelbine® Oral
  Arms: B
Drug: Carboplatin — Day 1: Carboplatin infusion AUC = 5 (Calvert's formula)
  Arms: B

SUMMARY:
The purpose of this study is to explore if the combination of vinorelbine and gemcitabine is better than vinorelbine and carboplatin in the treatment of advanced non-small cell lung cancer, in terms of survival, quality of life and need for palliative radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer stage IIIB or IV
* Not eligible for radical radiotherapy or surgery
* WHO performance status 0-2

Exclusion Criteria:

* Pregnancy
* Other clinical active cancer disease
* ALAT/ALP more than 3 times upper normal limit, bilirubin >1.5 upper limit
* Bowel disease that causes malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2007-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
survival | one year

SECONDARY OUTCOMES:
Health related quality of life (HrQoL) | 3 months
Toxicity | 3 months
Need for palliative radiotherapy | one year

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Fløtten, Study Chair — Haukeland University Hospital, thoracic department
Locations (4):
- Norway (4):
  - Øystein Fløtten, Bergen
  - Sverre Fluge, Haugesund
  - Heidi Rolke, Kristiansand
  - Tore Amundsen, Trondheim